CLINICAL TRIAL: NCT03969914
Title: PEEP-induced Changed in RRI as Physiological Background of Ventilator-induced Kidney Injury
Acronym: PRE-VIKI
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Alberto Fogagnolo, Principal investigator, Università degli Studi di Ferrara
Other Study IDs: RRIPEEP
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Respiratory Distress Syndrome, Adult; Respiration, Artificial; Acute Kidney Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill ventilated patients: Patients admitted to ICU with expected mechanical ventilation >48h
  Interventions: Procedure: PEEP changes

INTERVENTIONS:
Procedure: PEEP changes — All patients will be ventilated with a tidal volume of 6 ml/kg before the RRI assessment. Further, three level of PEEP (5, 10 and 15 cmH2O) will be randomly set. For each levels of PEEP, the RRI will be evaluated

SUMMARY:
The renal Doppler resistive index (RRI) is a noninvasive tool that has been used to assess renal perfusion in the intensive care unit (ICU) setting. Many parameters have been described as influential on the values of renal RI. Mechanical ventilation is associated with significant increases in the risk of acute kidney injury (AKI). Ventilator-induced kidney injury (VIKI) is believed to occur due to changes in hemodynamics that impair renal perfusion. The investigators hypothesized that patients who need mechanical ventilation should have a different response in RRI when different levels of Positive end expiratory pressure (PEEP) are applied. Investigators wish to describe changing in RRI due to changes in PEEP and to verify whether these changes could partially explain the occurrence of VIKI

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU with expected mechanical ventilation >48h

Exclusion Criteria:

* Ultrasound RRI evaluation non available
* Patients with arrhythmia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of critically ill patients
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Occurence of AKI | once a day until day 7
  AKI will be defined according to Kidney Disease: Improving Global Outcomes (KDIGO) criteria

SECONDARY OUTCOMES:
Change in RRI at different level of PEEP | One a day until day 5
  To compare median difference of RRI at PEEP 5 and PEEP 15 in patients who will develop (or not) AKI

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Università di Ferrara, Ferrara
  - Università di Siena, Siena

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared under reasonable request to the principal investigator
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Fogagnolo A, Grasso S, Morelli E, Murgolo F, Di Mussi R, Vetrugno L, La Rosa R, Volta CA, Spadaro S. Impact of positive end-expiratory pressure on renal resistive index in mechanical ventilated patients. J Clin Monit Comput. 2024 Oct;38(5):1145-1153. doi: 10.1007/s10877-024-01172-z. Epub 2024 May 21. PMID 38771490